CLINICAL TRIAL: NCT00509093
Title: A Phase 2 Study of Imatinib Mesylate (Gleevec) as Maintenance Therapy After Induction and Consolidation Chemotherapy in Patients With Newly Diagnosed C-kit Positive Acute Myeloid Leukemia
Brief Title: Imatinib Mesylate in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia Who Have Received Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4906; P30CA043703 (NIH); CASE4906 (Other: Case Comprehensive Cancer Center); AUS259 (Other: Novartis); NCI-2010-01198 (Other: NCI/CTRP)
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Leukemia
Keywords: adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myelomonocytic leukemia (M4); adult acute megakaryoblastic leukemia (M7); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult acute myeloid leukemia in remission
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute | interventions — Imatinib Mesylate; Gene Expression Profiling; Polymerase Chain Reaction; Flow Cytometry; Proto-Oncogene Proteins c-kit; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib Mesylate (Experimental)
  Interventions: Drug: imatinib mesylate; Genetic: gene expression analysis; Genetic: mutation analysis; Genetic: polymerase chain reaction; Other: flow cytometry; Procedure: biopsy

INTERVENTIONS:
Drug: imatinib mesylate — Patients will receive treatment with imatinib mesylate at a dose of 600 mg by mouth once a day for 12 months. The study dose can be split but the dose of 600 mg must be given within a 12 hour period.
  Other Names: Gleevec
Genetic: gene expression analysis — Multidrug resistance genes: These studies will include: MDR1, MRP1, LRP, and BCRP. Bone marrow blocks or cut slides will be sent to Duke on the diagnostic AML samples. DNA will be eluted from the samples so that the above genes can be analyzed.
  Other Names: MRD
Genetic: mutation analysis — FLT3 mutation analysis (on bone marrow aspirate or peripheral blood): These analyses will be performed by pathology at the time of diagnosis, at the participating institution. Samples will be analyzed for the FLT3 ITD and/or D835 mutation by PCR.
  Other Names: FLT3
Genetic: polymerase chain reaction — AF1q gene analysis (on bone marrow aspirate)
  Other Names: AF1Q gene analysis
Other: flow cytometry — C-kit MFI on AML samples will be calculated by using a CD45/ orthogonal light scatter gate to isolate blasts. The MFI will be calculated as the c-kit mean channel number (MCN) of the blasts/ MCN auto fluorescence.
  Other Names: C-kit MFI, CD117
Procedure: biopsy — Diagnostic bone marrow biopsy/aspirate must be done within 3 weeks of registration documenting complete remission
  Other Names: bone marrow biopsy/aspirate

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well imatinib mesylate works in treating patients with newly diagnosed acute myeloid leukemia who have received chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether adding imatinib mesylate as maintenance therapy improves progression-free survival in patients with c-kit positive acute myeloid leukemia (AML) compared with historical controls.

Secondary

* To assess the feasibility of administering imatinib mesylate as maintenance therapy after the completion of induction and consolidation therapy in these patients.
* To evaluate potential mechanisms of relapse/resistance in c-kit positive AML by examining multidrug resistance gene expression and AF1q gene expression and to determine whether these levels correlate with c-kit expression.

OUTLINE: This is a multicenter study.

Patients receive oral imatinib mesylate once daily for up to 12 months.

Bone marrow and peripheral blood are collected at baseline. Laboratory endpoints are evaluated by flow cytometry; mutation and gene analysis by PCR.

ELIGIBILITY:
INCLUSION CRITERIA

* Diagnostic bone marrow aspirate/ biopsy or peripheral blood confirming AML.
* At the time of diagnosis, patients must have c-kit (also known as CD117) positive AML (20% or more of the blasts express c-kit[CD117]).
* A flow scattergram (from the diagnostic AML specimen) must be available to calculate a c-kit MFI.
* Patients must have received standard induction chemotherapy with ADE (cytarabine, daunorubicin, and etoposide) or with 7+3 (7 days of cytarabine continuous infusion and 3 days of an anthracycline (idarubicin, daunorubicin, or mitoxantrone). Patients with persistent leukemia on a Day 10-28 marrow may have received a second course of chemotherapy.
* After the completion of induction therapy, patients must have attained a complete remission based on blood count recovery (neutrophil count ≥ 1,000/µL, platelet count ≥ 100,000/µL), and bone marrow aspirate and biopsy (< 5% myeloblasts).
* For patients < 60 years of age, patients must have received at least 2 courses of post-remission therapy with at least intermediate dose (400 mg/m2/day). *Patients with t(8;21) or inversion 16 at the time of diagnosis must have received at least 2 courses of high dose cytarabine. For patients > or = 60 years of age, patients must have received 1 course of post-remission therapy (the type of chemotherapy will not be specified).
* Patients must be registered on this study (maintenance Imatinib mesylate) within 60 days of the last dose of post-remission therapy.
* A bone marrow aspirate and/or biopsy must be done within 3 weeks of registration documenting CR.
* Women of childbearing potential and sexually active males must use an effective method of contraception.
* Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
* ECOG Performance Status 0-2.
* Creatinine must be ≤ 1.5 x upper limit of normal.
* Total bilirubin must be ≤ 2 mg/dl and AST and ALT must be ≤ 2 times the upper limit of normal.
* Previous treatment-related toxicities must have resolved to ≤ Grade 1 excluding alopecia.
* Written, voluntary informed consent.

EXCLUSION CRITERIA

* Acute promyelocytic leukemia.
* Patients with an autologous or allogeneic bone marrow transplant.
* History of HIV.
* Pregnant or breast-feeding.
* Serious or poorly controlled medical conditions that would interfere with the protocol.
* At the time of study entry, any medications which could significantly interact with imatinib mesylate must be discontinued.
* Patients with active extramedullary disease are not eligible.
* Patient has received any other investigational agents within 28 days of first day of study drug dosing.
* Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
* Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
* Patient previously received radiotherapy to ≥ 25 % of the bone marrow
* Patient had a major surgery within 2 weeks prior to study entry.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2014-05-09 (Actual); Study Completion 2015-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Brenda Cooper, MD, Principal Investigator — University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib Mesylate: Imatinib mesylate: Participants will receive treatment with imatinib mesylate at a dose of 600 mg by mouth once a day for 12 months. Study dose can be split but the dose of 600 mg must be given within a 12 hour period.
  Gene expression analysis: Multidrug resistance genes: These studies will include: MDR1, MRP1, LRP, and BCRP. Bone marrow blocks or cut slides will be sent to Duke on the diagnostic AML samples. DNA will be eluted from the samples so that the above genes can be analyzed.
  Mutation analysis: FLT3 mutation analysis (on bone marrow aspirate or peripheral blood): These analyses will be performed by pathology at the time of diagnosis, at the participating institution. Samples will be analyzed for the FLT3 ITD and/or D835 mutation by PCR.
  PCR: AF1q gene analysis (on bone marrow aspirate)
  Flow cytometry: C-kit MFI on AML samples will be calculated by using a CD45/ orthogonal light scatter gate to isolate blasts. The MFI will be calculated a
Period: Overall Study
Arm/Group | Imatinib Mesylate
Started | 32
Completed | 8
Not Completed | 24
Not completed — Adverse Event | 10
Not completed — Disease Progression | 9
Not completed — Transformed into MDS | 1
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (16.0)
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 4
  30-39 years | 3
  40-49 years | 4
  50-59 years | 10
  60-69 years | 4
  70-79 years | 6
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival (PFS) for Patients Less Than 60 Years of Age
Description: PFS measured from the date of Complete Response (CR) to the date of relapse or death. Progression defined as any of the following event: progression to accelerated phase or blast crisis, death, loss of CHR or MCyR, or in patients not achieving a CHR an increasing WBC despite appropriate therapeutic management
  This outcome will be reported as median progression-free survival in months for participants less than 60 years of age.
Time Frame: up to 5 years from the End of Treatment
Population: All participants less than 60 years of age
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 21
months | 52.1 [9.3 to NA] — Not enough events to estimate upper limit of 95% confidence interval

2. Primary Outcome: Progression-free Survival for Patients 60 Years of Age and Older
Description: Progression free survival will be measured from the date of Complete Response (CR) to the date of relapse or death.
Time Frame: up to 5 years from the End of Treatment
Population: All participants 60 years or older.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 11
months | 10.7 [1.7 to 20.8]

3. Primary Outcome: Percent of Participants Less Than 60 Years of Age With PFS at 8 and 13 Months Post-treatment
Description: Percent of participants less than 60 years of age with PFS at 8 and 13 months post-treatment
Time Frame: at 8 and 13 months after treatment.
Population: All participants less than 60 years of age
Measure: Number; unit: percent of participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 21
percent of participants
  at 8 months post treatment | 76.2
  at 13 months post treatment | 54.5

4. Primary Outcome: Percent of Participants 60 Years of Age or Older With PFS at 8 and 13 Months Post-treatment
Description: Percent of participants 60 years of age or older with PFS at 8 and 13 months post-treatment
Time Frame: at 8 and 13 months after treatment.
Population: All participants 60 years or older
Measure: Number; unit: percent of participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 11
percent of participants
  at 8 months post treatment | 61.9
  at 13 months post treatment | 36.4

5. Secondary Outcome: Toxicity as Measured by NCI CTC v. 3.0
Description: Number of patients (%) experiencing an adverse event
  See adverse events section for details
Time Frame: 13 months from start of treatment
Population: Number of patients (%) experiencing the adverse event
Measure: Count of Participants; unit: Participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 32
Participants | 30

6. Other Pre Specified Outcome: Correlation of C-kit Expression With Multidrug Resistance Gene Expression (MDR1, MRP1, LRP, and BCRP) and AF1q Expression
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to four weeks after off-study date, an average of 2.6 years
Arm/Group | Imatinib Mesylate
All-Cause Mortality (participants affected / at risk) | 20/32
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=32)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (2)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Infection with unknown ANC - Blood (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Pain - Bone (Nervous system disorders) | 1 (1)
Pain - Cardiac/heart (Nervous system disorders) | 1 (1)
Pain - Joint (Nervous system disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=32)
Fullness in Right Ear (Ear and labyrinth disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 12 (35)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 14 (41)
Lymphopenia (Blood and lymphatic system disorders) | 6 (47)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 14 (30)
Platelets (Blood and lymphatic system disorders) | 18 (53)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1 (2)
Hypotension (Cardiac disorders) | 1 (1)
aches at base of skull (General disorders) | 1 (1)
aural stuffiness (General disorders) | 1 (1)
body aches and chills (General disorders) | 1 (1)
Decreased total protein in blood (General disorders) | 1 (1)
Dyspnea (General disorders) | 1 (1)
edema in extremities (General disorders) | 1 (1)
emesis (General disorders) | 2 (2)
episode of flu (General disorders) | 1 (11)
facial edema (General disorders) | 1 (1)
facial itching (General disorders) | 1 (1)
hand stiffness (General disorders) | 1 (1)
Edema to face and legs (General disorders) | 1 (1)
Insomnia (General disorders) | 5 (5)
intermittent rash (General disorders) | 1 (1)
loose stool (General disorders) | 1 (1)
lower extremity edema (General disorders) | 1 (1)
mild edema in general and particularly in eye area (General disorders) | 1 (1)
mild swelling/edema (General disorders) | 1 (1)
mild tingling and discomfort rt lower extremity (General disorders) | 1 (1)
muscle cramping (General disorders) | 1 (1)
nasal congestion (General disorders) | 1 (1)
nausea (General disorders) | 2 (2)
occasional mild sore throat (General disorders) | 1 (1)
periorbital edema (General disorders) | 1 (1)
peri-orbital itchiness (General disorders) | 1 (1)
Periorbital swelling (General disorders) | 1 (1)
post nasal discharge (General disorders) | 1 (1)
post-herpetic neuralgia (General disorders) | 1 (1)
puffiness of eyes (General disorders) | 1 (1)
right heel pain (General disorders) | 1 (1)
right shoulder discomfort (General disorders) | 1 (1)
sore throat (General disorders) | 1 (1)
soreness in left ear (General disorders) | 1 (1)
stiff neck (General disorders) | 1 (1)
stomach burning (General disorders) | 1 (1)
upper back discomfort (General disorders) | 1 (1)
upper respiratory infection (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 13 (17)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Sweating (diaphoresis) (General disorders) | 1 (1)
Weight gain (General disorders) | 6 (6)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (General disorders) | 1 (1)
Dry skin (General disorders) | 1 (1)
blisters on feet (Skin and subcutaneous tissue disorders) | 1 (1)
discoloration of face (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (8)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 3 (5)
Anorexia (Skin and subcutaneous tissue disorders) | 2 (3)
Constipation (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 13 (20)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Upset Stomach (Gastrointestinal disorders) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 17 (30)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8)
Hemorrhage, GU - Urinary NOS (Gastrointestinal disorders) | 1 (1)
Infected cyst in left groin area; draining pus (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Renal and urinary disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Conjunctiva (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Nerve-peripheral (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1)
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1 (1)
Edema: head and neck (Infections and infestations) | 8 (9)
Edema: limb (Infections and infestations) | 12 (12)
Edema: trunk/genital (Blood and lymphatic system disorders) | 1 (1)
Edema: viscera (Blood and lymphatic system disorders) | 1 (1)
"Clear Liquid" coming from left ear (Blood and lymphatic system disorders) | 1 (1)
Small Preauricular Left Node (Blood and lymphatic system disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Blood and lymphatic system disorders) | 1 (1)
Alkaline phosphatase (Blood and lymphatic system disorders) | 4 (5)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4 (7)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 5 (7)
Bilirubin (hyperbilirubinemia) (Investigations) | 2 (3)
Calcium, serum-low (hypocalcemia) (Investigations) | 3 (5)
Creatinine (Investigations) | 2 (2)
Glucose, serum-high (hyperglycemia) (Investigations) | 4 (6)
Magnesium, serum-low (hypomagnesemia) (Investigations) | 1 (1)
Potassium, serum-high (hyperkalemia) (Investigations) | 1 (1)
Potassium, serum-low (hypokalemia) (Investigations) | 2 (2)
Sodium, serum-low (hyponatremia) (Investigations) | 3 (4)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extraocular (Investigations) | 1 (1)
Dizziness (Investigations) | 2 (2)
Neuropathy: sensory (Musculoskeletal and connective tissue disorders) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Mood alteration - Anxiety (Nervous system disorders) | 2 (2)
Mood alteration - Depression (Nervous system disorders) | 1 (1)
Eye Swelling and Redness (Psychiatric disorders) | 1 (1)
occasional burning of eyes (Psychiatric disorders) | 1 (1)
Optic disc edema (Eye disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Pain - Abdomen NOS (Eye disorders) | 4 (5)
Pain - Back (Eye disorders) | 1 (1)
Pain - Bone (Nervous system disorders) | 1 (1)
Pain - External ear (Nervous system disorders) | 1 (1)
Pain - Extremity-limb (Nervous system disorders) | 2 (2)
Pain - Head/headache (Nervous system disorders) | 3 (3)
Pain - Joint (Nervous system disorders) | 3 (3)
Pain - Muscle (Nervous system disorders) | 1 (1)
Mild Generalized Body Aches (Nervous system disorders) | 1 (1)
rt ankle pain (Nervous system disorders) | 1 (1)
chronic hip pain (Nervous system disorders) | 1 (1)
lower extremity pain (Nervous system disorders) | 1 (1)
mild cramping (Nervous system disorders) | 1 (1)
sciatica (Nervous system disorders) | 1 (2)
Pain - Pain NOS (Nervous system disorders) | 1 (1)
Pain - Stomach (Nervous system disorders) | 2 (6)
Pain - Throat/pharynx/larynx (Nervous system disorders) | 1 (1)
Bronchospasm, wheezing (Nervous system disorders) | 1 (1)
Cough (Nervous system disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased Bladder Pressure (Renal and urinary disorders) | 1 (1)
No Menstrual (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes